CLINICAL TRIAL: NCT06414070
Title: Jenga Dada: A Group-based Intervention to Prevent Partner Violence and Unintended Pregnancy Among Women in Kenya
Brief Title: Developing and Testing the Jenga Dada Intervention in Kenya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Population Council Kenya (Unknown); Women's Empowerment Link (Unknown); San Diego State University (Other)
Responsible Party: Principal Investigator, Jay G. Silverman, PhD, Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 800987
Record Dates: First submitted 2024-05-10; First posted 2024-05-16 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Reproductive Coercion; Intimate Partner Violence
Keywords: Reproductive coercion; Intimate partner violence; Contraceptive Use; Economic Abuse

STUDY DESIGN:
Intervention Model Description: Cluster-randomized controlled trial; stratified randomization based on urban/rural location
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Jenga Dada (Experimental): Jenga Dada programming in women's economic empowerment group meetings
  Interventions: Behavioral: Jenga Dada
- Waitlist Control (No Intervention): Standard women's economic empowerment group programming

INTERVENTIONS:
Behavioral: Jenga Dada — Jenga Dada aims to empower women participating in community-based economic groups by training them to recognize inequality, challenge it, and work toward positive changes in their lives related to finances, health, and relationships and increase social support on these issues within the groups. Jenga Dada is expected to include eight modules: 1) overview of the intervention, 2) gender roles, 3) economic control and abuse, 4) intimate partner violence (IPV), 5) reproductive coercion (RC), 6) family planning (FP), 7) financial literacy, and 8) life goals. The Jenga Dada intervention is group discussion-based and draws on two effective interventions: ARCHES (a facility-based contraceptive counseling intervention providing support for RC and IPV) and Girls Invest (a mobile health application with integrated modules on gender, IPV, and financial literacy). The intervention will be facilitated by a local NGO in partnership with group leaders.
  Arms: Jenga Dada

SUMMARY:
This study aims to work with women's economic empowerment groups within the community to address reproductive coercion and intimate partner violence and promote economic self-sufficiency among women (aged 15+ years). Based on the investigators' previous research in the United States, Bangladesh, and Kenya, the ARCHES (Addressing Reproductive Coercion in Health Settings) intervention is a highly effective clinic-based model to improve women's ability to use family planning and cope with abuse. Due to common requests for community-based support, content from the ARCHES intervention along with Girls Invest, an economic empowerment intervention implemented in the US and Nigeria, is being adapted to develop Jenga Dada, which means "Build a Woman Up" in Kiswahili, to be delivered to women's economic empowerment groups. The study will conduct formative research among women's economic empowerment group members, develop the Jenga Dada intervention, and conduct a pilot cluster randomized controlled trial to assess preliminary efficacy of the intervention on proximal outcomes (i.e., self-efficacy) and feasibility and acceptability.

DETAILED DESCRIPTION:
Background: This project aims to develop and preliminarily evaluate an intervention, Jenga Dada, on its feasibility, acceptability, and efficacy to increase women's and girl's ability to successfully cope with reproductive coercion (RC), intimate partner violence (IPV), economic abuse, and promote reproductive health and economic self-sufficiency among women participating in economic empowerment groups in rural and peri-urban areas of Uasin Gishu county, Kenya. Jenga Dada is being developed as an innovative hybrid approach based on adaptation and integration of core content from two effective interventions: ARCHES (Addressing Reproductive Coercion in Health Settings) and Girls Invest. ARCHES is a clinic-based contraceptive counseling intervention designed and demonstrated to support voluntary contraceptive use and reduce physical IPV. ARCHES was originally designed in the U.S. and has been adapted to and evaluated, with positive results, in Bangladesh and Nairobi, Kenya, and is currently being adapted for scale-up in public sector facilities in Uasin Gishu county, Kenya. Girls Invest is a mobile health application (mHealth app) with integrated intervention modules on gender, IPV, and financial literacy demonstrated to be feasible and acceptable among adolescent girls in the U.S. and Nigeria (efficacy evaluation ongoing). Jenga Dada combines the information and education from ARCHES and Girls Invest in a group discussion-based curriculum, delivered by a local women's empowerment non-governmental organization (NGO), that aims to build social support for women, delivered within women's economic empowerment groups as they move towards economic self-sufficiency, reproductive autonomy, and violence-free relationships.

Intervention: Jenga Dada educational sessions will be delivered to existing women's economic empowerment group participants during regular meetings by a facilitator from a local NGO. Sessions will include education and facilitated group discussions on gender, RC, IPV, economic abuse, and financial literacy to bolster understanding, shift attitudes and norms, and support peers on these issues. One 60-minute guided group discussion will take place for each of the eight training modules during the weekly or bi-weekly women's economic empowerment group meetings.

Methodology: This pilot trial will test the hypothesis that women participating in Jenga Dada will report improved proximal outcomes regarding a) coping with economic abuse, IPV, and RC (self-efficacy to seek assistance for IPV and coping strategies to maintain contraceptive use in the face of opposition) and b) self-efficacy to seek support for violence experiences from women's economic group members. Study activities include formative research to inform development of Jenga Dada based on the lived experience of women and girls and implementers in this context, pilot testing, and evaluation of the effects of Jenga Dada on violence, reproductive health, and economic outcomes. The evaluation will occur in two phases via random assignment of 18 existing women's economic empowerment groups to receive either Jenga Dada or standard women's economic empowerment group programming with baseline and 4-month follow-up survey data collected (n=280 participants, ages 15+ years). Post-program qualitative data from participants and implementers will be collected and analyzed to evaluate the feasibility and acceptability of the program.

ELIGIBILITY:
Inclusion Criteria:

* Being a women's economic group member prior to baseline
* Aged 15 years and older
* Able to provide informed consent
* Not planning to move out of the area or leave the women's economic group in the next 4 months

Exclusion Criteria:

* None

Min Age: 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Self-report biologically female
Enrollment: 279 (Actual)
Dates: Start 2024-06-17 (Actual); Primary Completion 2024-12-04 (Actual); Study Completion 2024-12-04 (Actual)

PRIMARY OUTCOMES:
Self-efficacy to cope with economic abuse | Baseline and 4-month follow-up
  Change in mean self-efficacy score (range: 6-18, higher=higher self-efficacy) between baseline and 4-month follow-up in intervention compared to control group (difference-in differences)
Self-efficacy to use family planning in the face of reproductive coercion among women of reproductive age (15-49 years) | Baseline and 4-month follow-up
  Change in mean self-efficacy score (range: 3-9, higher=higher self-efficacy) between baseline and 4-month follow-up in intervention compared to control group (difference-in differences)
Self-efficacy to seek formal intimate partner violence support services | Baseline and 4-month follow-up
  Change in mean self-efficacy score (range: 1-3, higher=higher self-efficacy) between baseline and 4-month follow-up in intervention compared to control group (difference-in differences)
Self-efficacy to seek support from the group/group members if experiencing violence (economic abuse, reproductive coercion among women of reproductive age [15-49 years], intimate partner violence) | Baseline and 4-month follow-up
  Change in mean self-efficacy score (range: 3-9 among women of reproductive age [15-49 years]; range: 2-6 for women above reproductive age [50+ years], higher=higher self-efficacy) between baseline and 4-month follow-up in intervention compared to control group (difference-in differences)

SECONDARY OUTCOMES:
Attitudes supportive of women's economic self-sufficiency | Baseline and 4-month follow-up
  Change in mean attitude score (range: 5-25, higher = more supportive attitudes) between baseline and 4-month follow-up in intervention compared to control group (difference-in differences)
Attitudes supportive of family planning use | Baseline and 4-month follow-up
  Change in mean attitude score (range: 7-35, higher = more supportive attitudes) between baseline and 4-month follow-up in intervention compared to control group (difference-in differences)
Attitudes not accepting of reproductive coercion | Baseline and 4-month follow-up
  Change in mean attitude score (range: 6-30, higher=attitudes less accepting of reproductive coercion/improved attitudes) between baseline and 4-month follow-up in intervention compared to control group (difference-in differences)
Attitudes not accepting of intimate partner violence | Baseline and 4-month follow-up
  Change in mean attitude score (range: 10-50, higher = attitudes less accepting of intimate partner violence/improved attitudes) between baseline and 4-month follow-up in intervention compared to control group (difference-in differences)
Awareness of intimate partner violence services | Baseline and 4-month follow-up
  Change in prevalence of awareness of intimate partner violence services between baseline and 4-month follow-up in intervention compared to control group (difference-in differences)
Family planning knowledge | Baseline and 4-month follow-up
  Change in mean knowledge score (range: 0-8, higher = more accurate knowledge) between baseline and 4-month follow-up in intervention compared to control group (difference-in differences)
Knowledge of financial resources | Baseline and 4-month follow-up
  Change in prevalence of knowledge of financial resources between baseline and 4-month follow-up in intervention compared to control group (difference-in differences)
Financial self-efficacy | Baseline and 4-month follow-up
  Change in mean self-efficacy score (range: 4-12, higher=higher self-efficacy) between baseline and 4-month follow-up in intervention compared to control group (difference-in differences)
Self-efficacy to access family planning services among women of reproductive age (15-49 years) | Baseline and 4-month follow-up
  Change in mean self-efficacy score (range: 4-12, higher=higher self-efficacy) between baseline and 4-month follow-up in intervention compared to control group (difference-in differences)
Self-efficacy to use a family planning method among women of reproductive age (15-49 years) | Baseline and 4-month follow-up
  Change in mean self-efficacy score (range: 4-12, higher=higher self-efficacy) between baseline and 4-month follow-up in intervention compared to control group (difference-in differences)
Self-efficacy to support someone experiencing violence (economic abuse, reproductive coercion, intimate partner violence) | Baseline and 4-month follow-up
  Change in mean self-efficacy score (range: 6-18, higher=higher self-efficacy) between baseline and 4-month follow-up in intervention compared to control group (difference-in differences)

OTHER OUTCOMES:
Group norms supportive of women's economic self-sufficiency | Baseline and 4-month follow-up
  Change in mean group norm score based off individual attitudes scales aggregated at group (i.e. cluster) level (range: 5-25, higher = more supportive norms) between baseline and 4-month follow-up in intervention compared to control group (difference-in differences)
Group norms supportive of family planning use | Baseline and 4-month follow-up
  Change in mean group norm score based off individual attitudes scales aggregated at group (i.e. cluster) level (range: 7-35, higher = more supportive norms) between baseline and 4-month follow-up in intervention compared to control group (difference-in differences)
Group norms not accepting of reproductive coercion | Baseline and 4-month follow-up
  Change in mean group norm score based off individual attitudes scales aggregated at group (i.e. cluster) level (range: 6-30, higher = norms less accepting of reproductive coercion/improved norms) between baseline and 4-month follow-up in intervention compared to control group (difference-in differences)
Group norms not accepting of intimate partner violence | Baseline and 4-month follow-up
  Change in mean group norm score based off individual attitudes scales aggregated at group (i.e. cluster) level (range: 10-50, higher = norms less accepting of intimate partner violence/improved norms) between baseline and 4-month follow-up in intervention compared to control group (difference-in differences)

CONTACTS AND LOCATIONS:
Overall Officials: Jay G Silverman, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- Community-based Women's Economic Empowerment Groups in Uasin Gishu County, Eldoret, Kenya

IPD SHARING:
Plan to Share IPD: Yes
Will share de-identified quantitative participant data analysis sets to the Dryad public data repository upon publication of findings
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Upon publication of findings
Access Criteria: Open access